CLINICAL TRIAL: NCT03707470
Title: The Effects of Made-To-Measure Compression Garments on Pressures Exerted on the Lower Limbs and Recovery From Muscle Damage in Rugby Players
Brief Title: Made to Measure Compression Garments for Recovery in Rugby Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St Mary's University College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMU_SHAS_2017_03
Record Dates: First submitted 2018-06-07; First posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Muscle Damage
Keywords: exercise induced muscle damage; recovery; rugby

STUDY DESIGN:
Intervention Model Description: Randomised, controlled, parallel trial
Who Masked: Participant
Masking Description: Participants to be provided with 2 different types of compression garments and a sham treatment (sham ultrasound) for recovery from muscle damaging exercise
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Custom fitted compression garments (CF) (Experimental): Custom fitted compression garments (Isobar, Manchester, UK) designed to provide 35 mmHg at the ankle and >20 mmHg at the mid-thigh (equivalent to European class 2 compression garments)
  Interventions: Device: Custom fitted compression garments (CF)
- Standard-sized compression garments (SSG) (Active Comparator): Off-the-shelf, standard-sized garments (2XU, Campbelltown, Australia), typically providing pressures equivalent to European grade 1 compression or below (5 - 15 mmHg at both the ankle and thigh)
  Interventions: Device: Standard-sized compression garments (SSG)
- Sham ultrasound (CON) (Sham Comparator): Sham ultrasound using an unplugged machine. Sham treatment for 5 minutes on each of the thighs, calves and hamstrings
  Interventions: Procedure: Sham ultrasound (CON)

INTERVENTIONS:
Device: Custom fitted compression garments (CF) — Custom fitted compression garments (Isobar, Manchester, UK) designed to provide 35 mmHg at the ankle and >20 mmHg at the mid-thigh (equivalent to European class 2 compression garments)
  Arms: Custom fitted compression garments (CF)
Device: Standard-sized compression garments (SSG) — Off-the-shelf, standard-sized garments (2XU, Campbelltown, Australia), typically providing pressures equivalent to European grade 1 compression or below (5 - 10 mmHg at both the ankle and thigh)
  Arms: Standard-sized compression garments (SSG)
Procedure: Sham ultrasound (CON) — Sham ultrasound using an unplugged machine. Sham treatment for 5 minutes on each of the thighs, calves and hamstrings
  Arms: Sham ultrasound (CON)

SUMMARY:
Aims

* To compare the compression pressures exerted by made-to-measure compression garments (CG) with those from standard sized garments
* To assess the efficacy of custom fitted, high pressure CG for facilitating the recovery of strength, muscular power and sprint performance, and to compare the effects with those of garments exerting lower pressures and a sham treatment

Rationale for study design

The results of a recent meta-analysis (unpublished data) have informed the design of this study. The conclusions of the meta-analysis were that CG are most effective for the recovery of:

* Force and power performance following eccentric/plyometric exercise
* Maximal force production, at least 24 hours post-exercise (for example in strength and power athletes undertaking resistance training programmes)
* Additionally, the recovery of high-intensity cardiovascular performance may also be enhanced by the used of CG, when tested 24 hours following exercise which incurs metabolic stress Accordingly, the current study was designed to investigate the effects of CG on the recovery of force, muscular power and sprint performance in rugby players over a 48 hour period following damaging exercise. The exercise protocol chosen (detailed below) provided both mechanical and metabolic recovery demands.

DETAILED DESCRIPTION:
Study 1) A comparison of the pressures exerted by different compression garments Participants were assessed for anthropometry; including height and body-mass, as well as waist, hip thigh, calf, ankle and gluteal circumferences. All limb measurements were taken from the right side, in accordance with guidelines set by the International Society of Anthropometry and Kinanthropometry (ISAK). Skinfold measurements were taken according to the ISAK 8 site protocol by a level 1 anthropometrist.

Thirty-two of the initially recruited 48 participants (see Study 2, below) were randomly selected and fitted for custom fitted compression garments (CG - stockings), after taking real-time 3D images using the manufacturer's proprietary, digitised method (Isobar, Manchester, UK). The custom fitted stockings (CF) were manufactured to apply pressures of 35 mmHg and 20 mmHg for the calf and mid-thigh respectively. Using a crossover design, applied pressures were compared to those from standard sized CG (SSG) which provided lower pressures (5-15 mmHg) for each athlete. Garments were provided in small, medium or large, dependent on athletes' size and fitted according to the manufacturer's guidelines based upon height and body-mass (2XU, Campbelltown, Australia). Pressures at the skin-garment interface were measured for both garments, worn in a randomised order, using a pressure monitor. Pressures applied at three sites were recorded: font-thigh and medial calf landmarks as defined by The International Society for the Advancement of Kinanthropometry (ISAK), and 2 cm above the centre of the median malleolus of the ankle. This visit to the laboratory took approximately 30 minutes per participant. Means and standard deviations were calculated from the pressure data to ascertain the average pressure exerted by the garments, as well as the variation in pressure across this population. Differences in measured pressures between garments were assessed using a paired-samples t-test (SPSS Statistics 22, IBM, New York, USA).

Study 2) An investigation into the effects of the pressures applied by different compression garments in facilitating the short term recovery of strength and power performance The full cohort of 48 athletes originally recruited participated in a randomised clinical trial (parallel design) to assess the effects of CG on recovery from a standardised eccentric exercise protocol. Athletes were required to avoid strenuous exercise for 48 hours before the start of the study, and then throughout 48 hours recovery. The first session included assessment of performance followed by a bout of damaging exercise and re-assessment, lasting approximately 90 minutes. Recovery was assessed in 2 further sessions, at 24 hours and at 48 hours after exercise (each lasting approximately 30 minutes).

Initial assessment Following a standardised warm up (400 m jogging, 20 leg swings in both the horizontal and sagittal planes on either leg, and any individual stretches usually performance by an athlete), maximal force production (using a strain-gauge - MIE Medical Research Ltd., Leeds, UK) was assessed by measuring the best of three attempts of maximal knee extension. Participants will be seated on a plyometric box, starting from a flexed position of 90o, as measured with a goniometer. In addition, 30 m sprint time (timing gates by Brower, Utah, USA) and vertical jump performance, using a jump mat (FSL electronics, Cookstown, UK), were assessed (best of 3 attempts). Soreness (200 mm visual analogue scale) and swelling (spring loaded tape measure - Lafayette Instrument Co, Lafayette, Indiana, USA) were also assessed. Muscle damage was also be quantified by creatine kinase analysis (RX Monza, Kearneysville, West Virginia, USA) from venous blood samples taken from the arm at baseline and at each time-point throughout recovery.

Eccentric muscle-damage protocol Following initial assessment, participants completed 20 sets of 20 m sprints with a 5 m deceleration phase, followed by 100 drop jumps. Sprints were separated by 60 s intervals. This combined protocol represents a novel and ecologically valid stimulus which combines the mechanical and metabolic stressors faced by Rugby Union players from competition and training. Sprints were timed to provide real-time feedback and encourage maximal effort, and sprints repeated if deceleration continued past the 5 m zone permitted. Subsequent drop jumps were performed from a 0.6 m platform, while athletes were encouraged to achieve the maximum height possible following a down-phase that resulted in the hips dropping below the level of the knee.

In a randomised, parallel-group design, athletes undertook either a sham treatment (CON), or wore CG immediately from the cessation of exercise for 48 hours recovery, removing them only to wash. Garments were manufactured to apply the pressures below, with no differences in physical appearance between garments. Athletes were allocated to one of the following three conditions:

* Custom fitted stockings (Isobar, Manchester, UK) applying over 35 mmHg and 20 mmHg at the calf and mid-thigh respectively (CF)
* Standard sized garments (2XU, Campbelltown, Australia) applying lower pressures (SSG - applying 5-15 mmHg, at both the calf and thigh)
* A sham ultrasound treatment (CON) The CON group received 15 minutes (5 minutes of quadriceps, 5 minutes of hamstrings, and 5 minutes of gastrocnemius) of sham ultrasound therapy (Combined therapy ultrasound/inferential; Shrewsbury Medical, Shropshire, United Kingdom) within 1 hour of the completion of performance testing. Pressures at the skin-garment interface were measured for both garments using a pressure monitor.

Performance measures - dependent variables Recovery was quantified by repeating the initial assessment and comparing to baseline values. Recovery of performance and recovery of markers of muscle damage were measured at the following time-points: pre-exercise, post-exercise, 24 hours post-exercise, 48 hours post-exercise. Between-group differences in the recovery of performance and physiological factors were assessed over time using a 2 way (time by condition) mixed-measures analysis of variance (SPSS Statistics 22, IBM, New York, USA).

All equipment used and methods employed made use of validated measures of strength, power, muscle damage and compression pressures.

ELIGIBILITY:
Inclusion Criteria:

* Actively playing
* A minimum of 2 years training experience.

Exclusion Criteria:

* Current injuries or illnesses
* Not actively playing at the time of testing
* Disruptions to training > 2 weeks within 8 weeks prior to testing

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change in lower body strength | Immediately post, 24 hours post, 48 hours post-exercise
  Change in maximal voluntary isometric contraction force of the knee extensors over time, measured in Newtons, using a force-meter to measure knee flexion force at 90 degrees
Change in lower body jump performance | Immediately post, 24 hours post, 48 hours post-exercise
  Change in maximal force from counter-movement jump over time, measured on a force platform (Newtons)
Change in sprint speed | Immediately post, 24 hours post, 48 hours post-exercise
  Change in 30 m sprint speed over time, measured using electronic timing gates

SECONDARY OUTCOMES:
Change in total haemoglobin concentration (tHb) | Immediately post-exercise, after having gone from the supine position (5 min), to standing (5 min)
  Accumulation of total haemoglobin, as measured with NIRS
Change in perceived soreness | Immediately post, 24 hours post, 48 hours post-exercise
  Change in perceived muscle soreness over time, measured by participants marking a line on a 200 mm visual analogue scale (from 0 mm - "no soreness"; to 200 mm - "worst soreness imaginable")
Change in creatine kinase concentrations (CK) | Immediately post, 24 hours post, 48 hours post-exercise
  Change in creatine kinase concentrations (IU) over time
Change in mid-thigh girth (MTG) | Immediately post, 24 hours post, 48 hours post-exercise
  Change in mid-thigh girth (cm) over time

CONTACTS AND LOCATIONS:
Locations (1):
- St Marys University, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Statistical Analysis Plan (SAP), Informed Consent Form (ICF), Clinical, Study Report (CSR) all available on request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Study Protocol, Statistical Analysis Plan (SAP), Informed Consent Form (ICF), Clinical, Study Report (CSR) all available on request from now until records are destroyed (after 10 years)
Access Criteria: Those requesting data should be planning a trial and provide their protocol, or be the participants whom the data belongs to

REFERENCES:
- [Background] Brophy-Williams N, Driller M, Halson S, Fell J, Shing C. Evaluating the Kikuhime pressure monitor for use with sports compression clothing. Sports Engineering. 2014;17(1):55-60.
- [Background] Jakeman JR, Byrne C, Eston RG. Lower limb compression garment improves recovery from exercise-induced muscle damage in young, active females. Eur J Appl Physiol. 2010 Aug;109(6):1137-44. doi: 10.1007/s00421-010-1464-0. Epub 2010 Apr 8. PMID 20376479
- [Background] Leeder J DC, van Someren KA, Gaze D, Jewell A, Deshmukh NI, Shah I, Barker J, Howatson G. Recovery and adaptation from repeated intermittent-sprint exercise. Int J Sports Physiol Perform. 2014 May;9(3):489-96. doi: 10.1123/ijspp.2012-0316. Epub 2013 Mar 8. PMID 23479406